CLINICAL TRIAL: NCT05608746
Title: Prehabilitation in Prostate Cancer Patients Undergoing Nerve Sparring Robot Assisted Radical Prostatectomy.
Brief Title: Prehabilitation in Prostate Cancer Patients, TelePrehabTrial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PREHABRHG001
Record Dates: First submitted 2022-10-25; First posted 2022-11-08 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise; Sex Counseling; Dietary Supplements

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Physical Exercise; Other: Pelvic Floor exercise; Other: Sexual counseling; Dietary Supplement: Nutritional supplement; Other: Stress management; Other: Standard pre-surgical preparation and pt. information.
- Control Group (Other)
  Interventions: Other: Standard pre-surgical preparation and pt. information.

INTERVENTIONS:
Other: Physical Exercise — Home-based individualized training, consisting of unsupervised aerobic exercise and resistance exercise, with moderate intensity. The pt. receives an exercise manual and exercise videos online, through an APP.
  Arms: Intervention Group
Other: Pelvic Floor exercise — Patients will be assessed by a physiotherapist and instructed in a pelvic floor exercise program, accessed through the APP. Furthermore, the pt. is provided with general information about pelvic floor anatomy and muscle function.
  Arms: Intervention Group
Other: Sexual counseling — Patients will be provided with 1 video-consultation with a clinical sexologist, during the prehabilitation period. The patients will be instructed in strategies to improve postoperative communication regarding, sex, realistic expectations, erectile dysfunction and the use of aids.
  Arms: Intervention Group
Dietary Supplement: Nutritional supplement — Patients are systematically screened for malnutrition to assess the nutritional status. Patients are given recommendations with dietary advice online, through the APP. If the patient is at nutritional risk, the patient is provided with a nutritional supplement.
  Arms: Intervention Group
Other: Stress management — Patients are systematically screened for anxiety and depression. If patients are at risk of anxiety or depression, they are referred to a consultation with a nurse, who will provide information and strategies to handle the uncertainties they may experience.
  Arms: Intervention Group
Other: Standard pre-surgical preparation and pt. information. — One week preoperatively the usual regime for the presurgical preparation and information will be followed.

SUMMARY:
Localized prostate cancer is commonly treated with radical prostatectomy (RP). Following surgery adverse effects such as urinary incontinence, erectile dysfunction associated with decreased quality of life and decreased physical function are common.

Traditionally, interventions to reduce these adverse effects are introduced postoperatively. However, a growing body of literature shows the benefit of interventions prior to surgery to enhance treatment success, known as prehabilitation.

Hence, the main purpose of this study is to develop and investigate the feasibility of prehabilitation using telehealth, to implement several interventions prior to elective RP.

ELIGIBILITY:
Inclusion Criteria:

* Male > 18 years
* Diagnosed with prostate cancer and referred to robot assisted nerve sparring RP
* Adequacy in written and spoken Danish
* Cognitively well-functioning
* Able to understand the study procedures and willing to provide signed informed consent

Exclusion Criteria:

* Severe comorbidities that would prevent the patient from exercising, e.g. recent fractures, severe heart disease or neurological disorders.
* No possibility to use a smartphone or tablet.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 12 months
  Percentage of eligible patients who accepted to participate in the study. Recruitment rate is measured by dividing the number of patients consented by the number of patients screened.
Protocol adherence, assessed by study-specific questionnaire | 12 months
  The pt. will every week register his adherence to the intervention protocol. The number of intervention components which were not fulfilled during the prehabilitation period will be counted, and the percentage of deviation will be calculated compared to the total number of intervention components.
Number of participants who received the nutritional and mental health intervention. | 12 months
  Total number of participants who after the initial screening, needed the Nutritional and Mental Health intervention.
Retention rate | 12 months
  Percentage of participants completing the full prehabilitation period, and full follow-up after the surgery. Retention rate is measured by dividing the number of patients completing the study with the number of patients consented.

SECONDARY OUTCOMES:
6-minute-walk-test (6MWT) | 12 months
  The 6MWT is a performance-based sub-maximal exercise test, used to assess aerobic capacity and endurance. The test covers the distance a person can walk on a 30-meters walkway, in the time of 6 minutes.
30 seconds sit-to-stand test (30STS) | 12 months
  30STS test is used to assess the leg strength and endurance. The test discovers how many times a person is able to rise up and sit down from a chair within 30 seconds.
Grip strength test | 12 months
  Grip strength is a measure of muscular strength or the maximum force/tension generated by the forearm muscles.
Self-reported physical activity | 12 months
  A questionnaire measuring physical activity consisting of three questions designed by The Swedish National Board of Health and Welfare (BHW).
Hospital Anxiety and Depression Scale (HADS) | 12 months
  Hospital Anxiety and Depression Scale is a questionnaire used to identify anxiety disorders and depression among patients in nonpsychiatric hospital clinics. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains.
12-Item short form Health Survey (SF-12) | 12 months
  The SF-12 is a short form of the 36-Item Short-form Health Survey (SF-36). It contains 12 items, and is a patient-reported survey of the patient's perception of health related quality of life, during the last 4 weeks.
5-Item International Index of Erectile Function (IIEF-5) | 12 months
  IIEF-5 is an abridged five-item version of the International Index of Erectile Function. It is a self-administered, multi-dimensional measure of erectile function.
24-hour Pad Weigh Test | 6, 24 and 50 weeks post surgery.
  The 24-hour Pad Weigh Test is used to investigate urinary incontinence.
Nutritional Risk Screening | At baseline (4 weeks before the surgery).
  NRS-2002 is a validated tool for nutritional screening of patients between 18 and 90 years of age.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Hospital Goedstrup, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No